CLINICAL TRIAL: NCT00562536
Title: Delayed Umbilical Cord Clamping in Infants Less Than 32 Weeks: A Randomized Controlled Trial
Brief Title: Delayed Umbilical Cord Clamping in Infants Less Than 32 Weeks
Acronym: DUC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mount Sinai Hospital Toronto
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Premature Birth
Keywords: Umbilical cord clamping; Preterm infants; Randomized controlled trial; For women giving birth to singleton infants 32 weeks gestational age or less
MeSH Terms: conditions — Premature Birth | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A 1 (Experimental): Delayed umbilical cord clamping 30-45 seconds.
  Interventions: Procedure: Umbilical cord clamping
- A 2 (No Intervention): Immediate umbilibcal cord clamping

INTERVENTIONS:
Procedure: Umbilical cord clamping — Delay of umbilical cord clamping 30 to 45 seconds
  Arms: A 1

SUMMARY:
The overall objective of the present study is to examine the effects of delayed umbilical cord clamping in preterm infants on neonatal outcomes using a prospective randomized controlled trial comparing immediate cord clamping (standard at present) with delayed cord clamping.

Our specific aim is to determine if a 30 to 45 second delay in umbilical cord clamping improves neonatal outcome as assessed by a composite of intraventricular hemorrhage and late onset sepsis in preterm infants born between 24 and 32 weeks gestation. Secondary outcomes to be examined include improvements in the following: 1) lung function as assessed by oxygen dependency at 36 weeks corrected gestational age (CGA), 2) cardiovascular function as assessed by the need for volume expansion, inotropes, or clinically suspected PDA requiring intervention prior to discharge home, and 3) anemia as assessed by initial hemoglobin, need for transfusion during stay in the NICU, and number of transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Women in labour or with a plan for delivery at a gestational age between 24 0/7 to 32 0/7 weeks gestation.
* Singleton pregnancy (Note: if pregnancy was a multiple gestation but demised occurred prior to 13 weeks, these patients can be included in study).

Exclusion Criteria:

* Moderate to life threatening fetal anomalies
* Multiple live gestations at birth (e.g. twins, triplets, etc)
* Intrauterine fetal demise
* Previous participation
* Stem cell collection

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 296 (Estimated)
Dates: Start 2007-11; Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Primary Composite outcome of Intraventricular Hemorrhage and/or Late Onset Sepsis | 3 years

SECONDARY OUTCOMES:
Secondary outcomes include: 1) lung function 2) cardiovascular function and 3) anemia. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kellie E Murphy, MD MSc, Principal Investigator — Mount Sinai Hospital, Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Chu KS, Shah PS, Whittle WL, Windrim R, Murphy KE. The "DUC" trial: a pilot randomized controlled trial of immediate versus delayed cord clamping in preterm infants born between 24 and 32 weeks gestation. J Matern Fetal Neonatal Med. 2021 Dec;34(24):4049-4052. doi: 10.1080/14767058.2019.1702959. Epub 2019 Dec 25. PMID 31875737